CLINICAL TRIAL: NCT04240483
Title: Intracutaneous Sterile Water Injections for Acute Low Back Pain in the Emergency Department: a Pilot Study
Brief Title: Intracutaneous Sterile Water Injections for Acute Low Back Pain in the Emergency Department
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study closed at Principal Investigator's request (study initiated, but not complete). Only 6 subjects had been recruited. The same study was just published.
Sponsor: Lindsey schmelzer (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Lindsey schmelzer, Principal Investigator, Mike O'Callaghan Military Hospital
Organization: Mike O'Callaghan Military Hospital (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FWH20200050H
Record Dates: First submitted 2020-01-21; First posted 2020-01-27 (Actual); Last update posted 2022-01-28 (Actual); Status verified 2022-01

CONDITIONS: Low Back Pain
Keywords: low back pain; sterile water injection; emergency department; sterile water; acute low back pain
MeSH Terms: conditions — Low Back Pain; Emergencies | interventions — Population Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intracutaneous sterile water injections (ISWI) group (Experimental)
  Interventions: Other: Intracutaneous sterile water injections (ISWI) group
- Intracutaneous dry injections (IDI) group (Sham Comparator)
  Interventions: Other: Intracutaneous dry injections (IDI) group

INTERVENTIONS:
Other: Intracutaneous sterile water injections (ISWI) group — ISWI consists of 4 intracutaneous injections of 0.5 ml sterile water in the lumbosacral region while patient is in a seated position. One injection given at the posterior superior iliac spine (Point 1) on both sides and second injection at 1 cm medial, and 1-2 cm inferior to the first point on both the sides (Point 2) using an insulin needle. These points overlie the area called Michaelis' rhomboid.
  Arms: Intracutaneous sterile water injections (ISWI) group
Other: Intracutaneous dry injections (IDI) group — Intracutaneous dry injections will be performed in the same manner described above, however, no sterile water or alternative solutions will be injected into the sites.
  Arms: Intracutaneous dry injections (IDI) group

SUMMARY:
The purpose of this study is to evaluate the efficacy of intracutaneous sterile water injections (ISWI) for treatment of acute low back pain in patients presenting to the emergency department. The primary aim is to determine if ISWI provides pain relief for acute low back pain in the ED. The secondary aim is to evaluate whether ISWI provides improved patient satisfaction in the ED setting. The hypothesis is that ISWI will improve pain amongst patients presenting with acute low back pain to the ED.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the efficacy of intracutaneous sterile water injections (ISWI) for treatment of acute low back pain in patients presenting to the emergency department. The primary aim is to determine if ISWI provides pain relief for acute low back pain in the ED. The secondary aim is to evaluate whether ISWI provides improved patient satisfaction in the ED setting. The hypothesis is that ISWI will improve pain amongst patients presenting with acute low back pain to the ED.

This pilot study will use a randomized controlled trial design to compare the effects of ISWI to intracutaneous dry injections in patients presenting to the ED with acute low back pain.

ELIGIBILITY:
**Patients must be able to get care at Nellis Air Force Base (a military installation) in order to participate in this study**

Inclusion Criteria:

* Active Duty and DoD Beneficiaries aged 18 to 64 years.
* Presenting to the ED with a chief complaint of acute low back pain of less than 2 weeks in duration.
* Pain severity on presentation of greater than or equal to 5/10 on Visual Analogue Scale.

Exclusion Criteria:

* Traumatic low back pain
* New weakness or neurologic deficit
* New loss bowel/bladder control
* Back pain above T12
* Active cancer
* Currently taking anticoagulant medications
* Signs of infection or trauma over the injection site
* Non-English speaking
* Pregnancy

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2020-07-27 (Actual); Primary Completion 2021-02-08 (Actual); Study Completion 2021-02-08 (Actual)

PRIMARY OUTCOMES:
Pain severity on 11-point Visual Analogue Scale (VAS) | pre-treatment
  Visual Analogue Scale (VAS) is a measurement instrument that tries to measure a characteristic or attitude that is believed to range across a continuum of values and cannot easily be directly measured.
  In this case the scale is accompanied by the Wong-Baker faces pain rating scale. Min pain score is 0, max pain score is 10. Lower scores mean a better outcome and higher scores mean greater pain severity.
Pain severity on 11-point Visual Analogue Scale (VAS) | 10 minutes post treatment
  Visual Analogue Scale (VAS) is a measurement instrument that tries to measure a characteristic or attitude that is believed to range across a continuum of values and cannot easily be directly measured.
  In this case the scale is accompanied by the Wong-Baker faces pain rating scale. Min pain score is 0, max pain score is 10. Lower scores mean a better outcome and higher scores mean greater pain severity.
Pain severity on 11-point Visual Analogue Scale (VAS) | 30 minutes post treatment
  Visual Analogue Scale (VAS) is a measurement instrument that tries to measure a characteristic or attitude that is believed to range across a continuum of values and cannot easily be directly measured.
  In this case the scale is accompanied by the Wong-Baker faces pain rating scale. Min pain score is 0, max pain score is 10. Lower scores mean a better outcome and higher scores mean greater pain severity.

SECONDARY OUTCOMES:
Satisfaction score on 11-point Visual Analogue Scale (VAS) | 30 minutes post treatment
  Visual Analogue Scale (VAS) is a measurement instrument that tries to measure a characteristic or attitude that is believed to range across a continuum of values and cannot easily be directly measured.
  In this case the VAS is a horizontal line ranging from left to right for unsatisfied to highly satisfied. Min pain score is 0, max pain score is 10.

CONTACTS AND LOCATIONS:
Overall Officials: Paul F Crawford, MD, Study Director — United States Air Force
Locations (1):
- Mike O'Callaghan Military Medical Center, Nellis Air Force Base, Nevada, United States

IPD SHARING:
Plan to Share IPD: No
We do not plan on sharing data

REFERENCES:
- [Background] Byrn C, Olsson I, Falkheden L, Lindh M, Hosterey U, Fogelberg M, Linder LE, Bunketorp O. Subcutaneous sterile water injections for chronic neck and shoulder pain following whiplash injuries. Lancet. 1993 Feb 20;341(8843):449-52. doi: 10.1016/0140-6736(93)90204-t. PMID 8094485
- [Background] Cui JZ, Geng ZS, Zhang YH, Feng JY, Zhu P, Zhang XB. Effects of intracutaneous injections of sterile water in patients with acute low back pain: a randomized, controlled, clinical trial. Braz J Med Biol Res. 2016 Mar;49(3):e5092. doi: 10.1590/1414-431X20155092. Epub 2016 Feb 2. PMID 26840703
- [Background] Genc Koyucu R, Demirci N, Ender Yumru A, Salman S, Ayanoglu YT, Tosun Y, Tayfur C. Effects of Intradermal Sterile Water Injections in Women with Low Back Pain in Labor: A Randomized, Controlled, Clinical Trial. Balkan Med J. 2018 Mar 15;35(2):148-154. doi: 10.4274/balkanmedj.2016.0879. Epub 2017 Oct 26. PMID 29072177
- [Background] Hosseininejad SM, Emami Zeydi A. Can intracutaneous sterile water injection be used as a possible treatment for acute renal colic pain in the emergency department? A short literature review. Urol Ann. 2015 Jan-Mar;7(1):130-2. doi: 10.4103/0974-7796.148669. No abstract available. PMID 25657569
- [Background] Martensson LB, Hutton EK, Lee N, Kildea S, Gao Y, Bergh I. Sterile water injections for childbirth pain: An evidenced based guide to practice. Women Birth. 2018 Oct;31(5):380-385. doi: 10.1016/j.wombi.2017.12.001. Epub 2017 Dec 11. PMID 29241699
- [Background] S, Valarmathy, and Josephine Hema j. "Intracutaneous sterile water injection over sacrum for the relief of low back pain in labour." Journal of Evolution of Medical and Dental Sciences, vol. 7, no. 28, 2018, pp. 3151-54, doi:10.14260/jemds/2018/709
- [Background] Skinner, Virginia, et al. "Sterile Water Injections for Relief of Back Pain in Labour - a Qualitative Study." Women and Birth, vol. 31, Oct. 2018, p. S50. ScienceDirect, doi:10.1016/j.wombi.2018.08.149
- See also: sterile water injections for pain relief — https://sciencebasedmedicine.org/sterile-water-injections-for-pain-relief/

DOCUMENTS (1):
  • Informed Consent Form (2020-03-24): https://cdn.clinicaltrials.gov/large-docs/83/NCT04240483/ICF_000.pdf